CLINICAL TRIAL: NCT07200726
Title: The Role of Neuroinflammation on Neurocognitive Outcome in Cardiac Surgery: INOCS Study
Brief Title: The Role of Neuroinflammation on Neurocognitive Outcome in Cardiac Surgery
Acronym: INOCS
Status: Recruiting | Type: Observational
Sponsor: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Sponsor
Other Study IDs: Z-2025013
Record Dates: First submitted 2025-09-05; First posted 2025-10-01 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-07

CONDITIONS: Postoperative Neurocognitive Dysfunction; Postoperative Neurocognitive Disorder; Cardiac Surgery; Major Surgery Under General Anesthesia; Major Surgery in Adult Patients; Postoperative Fatigue; Elderly Patients; Quality of Recovery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational study design - no intervention — Observational study design - no intervention

SUMMARY:
RATIONALE: Postoperative cognitive changes are common after cardiac surgery and can be categorised into three main types: postoperative delirium (POD), delayed neurocognitive recovery (DNCR) and postoperative neurocognitive disorder (PNCD). DNCR is diagnosed until postoperative day 30 and PNCD is diagnosed at least 30 days after the operation. Both conditions can be mild or major, and can affect the quality of life of these patients.

The incidence of PNCD in cardiac surgery is around 40%. Despite this high incidence, screening for PNCD is absent in current postoperative care since the diagnosis of PNCD is difficult and very time intensive. Furthermore, the underlying pathogenesis is incompletely understood.

The identification of a biomarker and/or validated short diagnostic instrument would be of paramount importance to easily identify patients at risk, or to diagnose patients with PNCD in order to identify therapeutical pathways for this disease.

OBJECTIVES: The main objective of this prospective clinical trial is to evaluate the performance of the short NPA and/or biochemical markers for the diagnosis of DNCR and PNCD in cardiac surgery patients aged 60 years or older.

STUDY DESIGN: Single-centre interventional observational study

STUDY INTERVENTIONS: Patients will undergo a neurophysiological assessment (NPA) pre-operatively and at two timepoints post-operatively, namely 6 (+/-1) days and 40 (+/- 10) days after surgery. During the stay at the intensive care unit, they will be screened daily for delirium, using the CAM-ICU and 3D-CAM.

To evaluate whether the development of DNCR or POD has an important effect on quality of recovery , the quality of recovery scale 15 (QOR-15), muscle strength (handgrip strength) and the Chalder fatigue score will be scored post-operative (postop day 1, 3 and 5). To evaluate whether PNCD has an effect on quality of live the EQ5D5L score will be measured at 40 (+/- 10) days after surgery, compared to preoperative values.

On several time points, blood samples will be drawn to measure markers of neuroinflammation. The time points will be preoperatively, at the moment of arrival on ICU, postoperative day 1, 2 and 3, if still on ICU. Two repeat blood sample will be taken at the moment of NPA performed after 6 (+/- 1) days and 40 (+/- 10) days after surgery, if the patient is willing (not obligatory).

STUDY POPULATION:

Patients aged 60 years or older who are scheduled for cardiac surgery.

Inclusion criteria:

* aged 60 years or older;
* scheduled for cardiac surgery.

Exclusion criteria:

* dementia, as diagnosed by a neurologist;
* urgent, not elective surgery.

MAIN STUDY ENDPOINTS:

Primary outcome PNCD defined as a decline of > 1 SD on > 2 tests in one or more cognitive domains or a decline of > 1 SD on total cognitive domain score.

Secondary outcomes Postoperative delirium - CAM-ICU will be evaluated twice daily (morning and evening) on every day when the patient is awake (not intubated) on the ICU. This is standard of care and is part of the routine clinical care in the hospital. Furthermore, once daily a 3D-CAM will be performed on day 1, 3 and 5.

Quality of recovery

* QOR-15, a validated measurement of quality of recovery in the short term postoperative recovery, will be evaluated pre-operatively and postoperatively day 1, 3 and 5.
* EQ5D5L, a validated measurement of quality of recovery in the long term postoperative recovery, will be evaluated preoperatively and at the moment of the third NPA measurement.
* Postoperative muscle function (upper extremity, by hand grip strength) on day 1, 3 and 5 after surgery and at the moment of the second and third NPA measurement (being day 6 (+/-1) and day 40 (+/-10) postoperatively), as compared to preoperative values.
* Chalder Fatigue questionnaire on day 1, 3 and day 5 and on the second and third NPA measurement, as compared to preoperative.

Biochemical analysis

- Blood samples will be drawn for analysis before induction of anaesthesia (preoperatively), at the end of the operation (immediately postoperatively on arrival in ICU), on day 1, 2 and 3 postoperatively (if still at the ICU) and at the time of the postoperative follow-up visits with the NPA testing (day 6 (+/-1) and day 40 (+/-10) days post-surgery).

At each time point, markers of neuroinflammation and -degeneration will be determined.

Tertiary outcomes

* Length of CPB
* Duration of mechanical ventilation
* Administered anaesthetic drugs during surgery
* Transfusion need
* Length of ICU stay (days)
* Length of in-hospital stay (days)
* Readmission to ICU or hospital within 28 days after surgery
* Cardiovascular outcome: atrial fibrillation, , thrombo-embolic events, myocardial injury, myocardial infarction, cardiac arrest, cardiac death
* Pulmonary outcome: postoperative pulmonary complications, postoperative pneumonia, postoperative respiratory failure
* Postoperative infection within 28 days after surgery

ELIGIBILITY:
Inclusion Criteria:

* aged 60 years or older;
* scheduled for cardiac surgery.

Exclusion Criteria:

* dementia, as diagnosed by a specialist, since this would make detection of PNCD impossible;
* urgent, not elective surgery.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Since, compared to younger patients undergoing major surgery, elderly patients are more prone to develop PNCD and are at greater risk of morbidity, we will therefore include patients aged 60 years or older scheduled for cardiac surgery.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-10-21 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative neurocognitive disorder (PNCD) after cardiac surgery using the NPA. | The NPA will be taken preoperatively and postoperatively on day 40 (+/- 10).
  The neuropsychological assessment (NPA) consists of 17 subsets which can be divided into five cognitive domains: speed and attention, memory, language, executive and visuospatial functioning. The outcomes are 21 scores, namely the scores of the 17 subsets and 4 combined scores. These are reported in T-scores after correction for age and educational level by comparison with a norm group. PNCD is defined as a decline of > 1 SD on > 2 tests in one or more cognitive domains or a decline of > 1 SD on total cognitive domain score.

SECONDARY OUTCOMES:
Delayed neurocognitive recovery (DNCR) | Day 6 (+/- 1) following surgery.
  Neurocognitive disorder early after surgery (< 30 days) will be assessed using the NPA (similar to the primary outcome).
Postoperative delirium (CAM-ICU) | Twice daily (morning and evening) day 1 - day 5 following surgery if the patient is still in the ICU.
  To assess postoperative delirium on the ICU the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) questionnaire will be done twice daily (morning and evening) every day when the patient is in the ICU. The CAM-ICU is a structured assessment tool. Based on the patient's responses and performance, it is determined whether delirium is present or not.
Postoperative delirium (3D-CAM) | Postoperative day 1, day 3 and day 5.
  To assess postoperative delirium the 3 minute confusion assessment method (3D-CAM) questionnaire will be done on day 1, day 3 and day 5 postoperatively. The 3D-CAM consists of a structured interview and cognitive testing. Based on the patient's responses and performance, it is determined whether delirium is present or not.
Quality of recovery (QoR-15) | Preoperative, postoperative day 1, day 3 and day 5.
  Quality of Recovery Score (QoR-15 score) is a patient-reported outcome measurement which will be used to assess the early postoperative health status of the patient after surgery and anaesthesia, i.e. the quality of recovery. The score is arbitrary and ranges from 0 to 150, the higher the score the better the quality of recovery.
Postoperative muscle strength (HGS) | Preoperative, postoperative day 1, day 3, day 5, day 6 (+/- 1), and day 40 (+/- 10).
  Postoperative muscle strength (upper extrimity) will be assessed by comparing the handgrip strength (HGS) of the dominant hand, measured on day 1, day 3, day 5, day 6 (+/- 1), and day 40 (+/- 10) following surgery as compared to the preoperative value.
Postoperative fatigue (CFQ) | Preoperative, postoperative day 1, day 3, day 5, day 6 (+/- 1), and day 40 (+/- 10).
  To assess general fatigue a fatigue questionnaire, the Chalder fatigue questionnaire (CFQ), will be taken on day 1, day 3, day 4, day 6 (+/- 1) and day 40 (+/- 10) postoperatively. The questionnaire consists of 11 items that assess both physical and mental aspects of fatigue. Respondents rate each item ranging from 0 to 3, the scores are then totaled to provide a measure of overall fatigue, a higher score meaning more severe fatigue.
Health-related quality of life (EQ5D5L) | Preoperative and postoperative day 40 (+/- 10).
  The EQ-5D-5L is used for measuring health-related quality of life. EQ-5D-5L provides a simple descriptive profile and a single index value for health status, both can be used to assess overall helaht. The descriptive profile consists of five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels of severity: no problems, slight problems, moderate problems, severe problems, or not able. Respondents select the level that best describes their current health status. The EQ-5D-5L also includes a visual analog scale (VAS) where respondents rate their current health status on a scale from 0 to 100, with 0 being the worst imaginable health state and 100 being the best imaginable health state.
Subjective sleep quality (PSQI) | Preoperative, postoperative day 6 (+/- 1), and day 40 (+/- 10).
  To assess subjective sleep quality the Pittsburgh Sleep Quality Index (PSQI) will be used. The PSQI consists of 19 items that assess different components of sleep, including sleep latency, sleep duration, sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction due to poor sleep quality. Each item is rated on a scale from 0 to 3, with higher scores indicating worse sleep quality. The scores from all 19 items are summed to provide a total score ranging from 0 tot 21, with higher scores indicating poorer sleep quality. The questionnaire will be filled in 3 times: before surgery, day 6 (+/-1) and day 40 (+/- 10) after surgery.
Sleeping EEG pattern | First postoperative night.
  Electroencephalographic (EEG) readings will be conducted during the first postoperative night to asses sleep architecture.
Markers of neuroinflammation and neurodegeneration | Before induction of anaesthesia, immediately postoperative (on arrival in ICU), day 1, day 2 and day 3 postoperative (if still in ICU), day 6 (+/- 1) and day 40 (+/- 10).
  Blood samples will be drawn for analysis before induction of anaesthesia (preoperatively), at the end of surgery on arrival in ICU, on day 1, 2 and 3 postoperatively (if still in the ICU) and at the time of follow-up visits on day 6 (+/- 1) and day 40 (+/- 10) post-surgery. Markers of neuroinflammation and neurodegeneration (Phospho-Tau, NfL) will be determined.

CONTACTS AND LOCATIONS:
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: No